CLINICAL TRIAL: NCT05289986
Title: Switch from Stable CART Containing ABA/3TC or TAF/FTC Plus Dolutegravir or Bictegravir to TDF/3TC/doravirine in People Living with HIV: Impact on Lipids, Body Composition, Insulin Sensitivity, Neuroendocrine Function and Inflammation Markers
Brief Title: The Effect on Lipid Profile of Switching to Delstrigo in HIV Positive Patients
Acronym: META-D
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The CI, sponsor and funder jointly made the decision to end the trial due to lack of recruitment, as well as due to delays it was felt value of the primary endpoint had lessened to a point where its scientific value was questioned.
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRF006
Record Dates: First submitted 2022-01-26; First posted 2022-03-22 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate switch arm (Experimental): Experimental arm (baseline visit switch group, N=30): One DOR/TDF/3TC tablet taken orally once daily for 48 weeks.
  Virally suppressed participants on a stable combined ART regimen will be randomised (1:1) to an immediate switch to 3TC/TDF/DOR (immediate switch arm, N=30) for the duration of the 48-week study, or to maintaining their current cART followed by a switch to 3TC/TDF/DOR from week 24-48 (delayed switch arm, N=30). Participants will be monitored for the length of the study (48 weeks) plus a 30-day follow-up period.
  Interventions: Drug: DELSTRIGO 100Mg-300Mg-300Mg Tablet
- delayed switch arm (Active Comparator): Control arm (deferred switch group, N=30): Participants will continue their current triple cART regimen for 24 weeks, and then switched to taking one TDF/3TC/DOR tablet orally once daily (24 -48 weeks).
  Virally suppressed participants on a stable combined ART regimen will be randomised (1:1) to an immediate switch to 3TC/TDF/DOR (immediate switch arm, N=30) for the duration of the 48-week study, or to maintaining their current cART followed by a switch to 3TC/TDF/DOR from week 24-48 (delayed switch arm, N=30). Participants will be monitored for the length of the study (48 weeks) plus a 30-day follow-up period.
  Interventions: Drug: DELSTRIGO 100Mg-300Mg-300Mg Tablet

INTERVENTIONS:
Drug: DELSTRIGO 100Mg-300Mg-300Mg Tablet — Delstrigo (300 mg of tenofovir disoproxil fumarate equivalent to 245 mg of tenofovir disoproxil, 300 mg of lamivudine and 100 mg of doravirine
  - TDF/3TC/DOR)

SUMMARY:
This is an open label, randomised, two-arm switch study over 48 weeks in which virally suppressed participants on a stable combined ART regimen will be randomised (1:1) to an immediate switch to 3TC/TDF/DOR (immediate switch arm, N=30) for the duration of the 48-week study, or to maintaining their current cART followed by a switch to 3TC/TDF/DOR from week 24-48 (delayed switch arm, N=30). Participants will be monitored for the length of the study (48 weeks) plus a 30-day follow-up period.

If patients withdraw or are withdrawn from the study treatment prematurely, an early termination visit (ETV) should occur within 30 days post withdrawal.

The hypothesis of the study is that a switch to Delstrigo, which is a combination of tenofovir disoproxil, lamivudine and doravirine (TDF/3TC/DOR) has a favourable impact on lipid metabolism, glucose, weight, body composition and hepatic steatosis.

DETAILED DESCRIPTION:
Open-label, 2 arm, multi-centre, non-inferiority switch study.

Sample size: 60 participants

Participant population: HIV-1 infected patients on stable and suppressive triple cART.

IMP: Delstrigo (300 mg of tenofovir disoproxil fumarate equivalent to 245 mg of tenofovir disoproxil, 300 mg of lamivudine and 100 mg of doravirine

- TDF/3TC/DOR)

Study setting: Patients will be identified through HIV clinic visits by their direct study medical care team and visits will be captured on a participant-screening log. A Trial Management Team will facilitate the project and liaise with participating sites in study set-up and progress.

Dose and Route of Administration:

Experimental arm (baseline visit switch group, N=30): One DOR/TDF/3TC tablet taken orally once daily for 48 weeks.

Control arm (deferred switch group, N=30): Participants will continue their current triple cART regimen for 24 weeks, and then switched to taking one TDF/3TC/DOR tablet orally once daily (24 -48 weeks).

Primary Objective To quantify the effect on lipid profile (change from baseline in total fasting cholesterol to Week 24) of switching from suppressive, stable cART containing ABA/3TC or TAF/FTC plus dolutegravir or bictegravir to Delstrigo (TDF/3TC/DOR) in HIV positive patients.

Secondary Objectives

To investigate the effect of switch on:

1. Body composition changes when measured by Total Body DXA at week 24 and 48 and by waist circumference
2. Change in insulin sensitivity from baseline to week 24 and 48 by HOMA-IR (glucose & insulin levels)
3. PBMC cholesterol and cholesteryl levels
4. Adipocytokines by assessing adiponectin, leptin
5. Pituitary hormones (TSH, LH, FSH, IGF-1, Testosterone)
6. Estimated cardiovascular risk (QRISK3 and D:A:D equations)
7. Hepatic steatosis and fibrosis by transient elastography-CAP (FibroScan® with the CAP probe)
8. Dietary, Quality of Life (EuroQoL), and Sleep quality (Pittsburgh Sleep Quality Index) Questionnaires
9. Renal safety by uPCR, eGFR Potential Exploratory Objectives Platelet aggregation & endothelial markers, metabolomics

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected, 18 years or older
* On stable & suppressive triple cART containing ABA/3TC or TAF/FTC plus dolutegravir or bictegravir for at least 6 months
* No evidence of resistance to TDF, 3TC, or DOR
* No laboratory abnormalities, medical/psychiatric conditions or alcohol/drug use considered a barrier to participation by investigators
* Women who are of childbearing potential and sexually active need to use the hormonal contraceptive methods, associated with inhibition of ovulation, listed in the protocol:

  * Implant
  * Depot injection
  * Intra-uterine device or system
  * Oral hormonal contraception A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
* Men who are sexually active and have partners who are women of childbearing potential must be using an adequate method of contraception to avoid pregnancy (male condom or sterilisation confirmed prior to the subject's entry into the study)

Exclusion Criteria:

* History of virological failure on an NNRTI in absence of a post-failure genotypic resistance test proving absence of resistance to DOR
* Concomitant medication contra-indicated with TDF, FTC or DOR
* Haemoglobin <9 g/dL
* Platelets <80,000/mm3
* Creatinine clearance <50 mL/min
* AST or ALT ≥5N
* Acute Hepatitis A infection.
* Concomitant DAA for anti-HCV therapy
* Known acute or chronic viral hepatitis B or C.

  o Individuals with positive anti-HCV results, but with HCV RNA not detected may be included on the trial.
* Pregnant or breastfeeding women, or individuals actively trying to conceive
* History of osteoporosis or bone fractures/loss
* Hypersensitivity to the active substance or to any of the excipients in tenofovir disoproxil fumarate, lamivudine and/or doravirine formulations
* Patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
To quantify the effect on lipid profile | 24 weeks
  To quantify the effect on lipid profile (change from baseline in total fasting cholesterol to Week 24) of switching from suppressive, stable cART containing ABA/3TC or TAF/FTC plus dolutegravir or bictegravir to Delstrigo (TDF/3TC/DOR) in HIV positive patients.

SECONDARY OUTCOMES:
Percentage of patients with treatment-related adverse events by week 48 | 48 weeks
  Percentage of patients with treatment-related adverse events by week 48
Median change in body fat content (g) measured by Total body dexa at week 24 and 48 | 48 weeks
  Median change in body fat content (g) measured by Total body dexa at week 24 and 48
Body composition changes when measured by waist circumference at week 24 and 48 | 48 weeks
  Body composition changes when measured by waist circumference at week 24 and 48
Change in insulin sensitivity from baseline to week 24 and 48 by HOMA-IR (glucose & insulin levels) | 48 weeks
  HOMA-IR is calculated by glucose & insulin levels and provides a single unit of measure
PBMC cholesterol and cholesteryl levels | 48 weeks
  PBMC cholesterol and cholesteryl levels
Adipocytokines by assessing adiponectin, leptin | 48 weeks
  Adipocytokines by assessing adiponectin, leptin
Pituitary hormones (TSH, LH, FSH, IGF-1, Testosterone) | 48 weeks
  Pituitary hormones (TSH, LH, FSH, IGF-1, Testosterone)
Estimated cardiovascular risk (QRISK3 equation) | 48 weeks
  Estimated cardiovascular risk (QRISK3 equation)
Estimated cardiovascular risk (D:A:D equation) | 48 weeks
  Estimated cardiovascular risk (D:A:D equation)
Hepatic steatosis and fibrosis by transient elastography-CAP (FibroScan® with the CAP probe) | 48 weeks
  Hepatic steatosis and fibrosis by transient elastography-CAP (FibroScan® with the CAP probe)
Dietary preferences (using Food preference questionnaire for adolescents and adults) | 48 weeks
  Dietary preferences (using Food preference questionnaire for adolescents and adults)
Quality of Life (EuroQoL questionnaire) | 48 weeks
  Quality of Life (EuroQoL questionnaire)
Sleep quality (Pittsburgh Sleep Quality Index questionnaire) | 48 weeks
  Sleep quality (Pittsburgh Sleep Quality Index questionnaire)
Renal safety by uPCR | 48 weeks
  Renal safety by uPCR
Renal safety by eGFR | 48 weeks
  Renal safety by eGFR

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital NHS Foundation Trust, London, London
  - Mortimer Market Centres, London, London

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will be provided reasonable access to statistical tables, figures, and relevant reports.
  Sponsor will also provide the investigators with the full summary of the study results. The investigator is encouraged to share the summary results with the study subjects, as appropriate.
  The procedures and timing for public disclosure of the results summary and for development of a manuscript for publication will be in accordance with sponsor policies.